CLINICAL TRIAL: NCT03856944
Title: Evaluating Refractive and Visual Outcomes With the Alcon Toric ReSTOR +2.5 and +3.0 Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gainesville Eye Associates (Other)
Collaborators: SiV Consulting (Other)
Responsible Party: Principal Investigator, Clayton Blehm, MD, Principal investigator, Gainesville Eye Associates
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CB-18-001
Record Dates: First submitted 2018-10-04; First posted 2019-02-27 (Actual); Results first posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: Cataract
Keywords: Astigmatism; intraocular lens; multifocal
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Intervention Model Description: This study is a prospective, single center, open clinical trial to collect normative performance data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- ReSTOR Toric (Experimental): Patients will be bilaterally implanted, with the Toric ReSTOR +2.5D model implanted in the dominant eye and the Toric ReSTOR +3.0D model implanted in the non-dominant eye. Patients will self-select for multifocal implantation.
  Interventions: Device: ReSTOR Toric

INTERVENTIONS:
Device: ReSTOR Toric — ReSTOR Toric bilateral IOL implantation
  Other Names: ReSTOR +2.5 Toric; ReSTOR +3.0 Toric

SUMMARY:
The study will evaluate visual acuity and visual function with a 'blended' ReSTOR Toric intraocular lens (IOL) implantation after cataract surgery.

DETAILED DESCRIPTION:
The objective is to provide a normative standard for refractive and visual outcomes in eyes with significant corneal astigmatism undergoing cataract surgery with the Alcon Toric ReSTOR lens. Patients will be bilaterally implanted, with the Toric ReSTOR +2.5D model implanted in the dominant eye and the Toric ReSTOR +3.0D model implanted in the non-dominant eye.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in the eligible eye.

* Bilateral visually-significant cataracts
* Willing and able to provide written informed consent for participation in the study.
* Willing and able to comply with scheduled visits and other study procedures.
* have good ocular health, with no pathology that compromises visual acuity (outside of residual refractive error and cataract)
* Regular corneal astigmatism of 1.00D to 2.50D in both eyes
* Potential postoperative acuity of 20/25 or better

Exclusion Criteria:

* If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

  * Irregular astigmatism (e.g. keratoconus)
  * Corneal pathology (e.g. opacities, epithelial basement membrane dystrophy (EBMD), Fuch's dystrophy, etc.)
  * Monocular status (e.g. amblyopia)
  * Previous radial keratotomy, corneal refractive surgery or other corneal surgery (e.g. corneal transplant, Descemet Stripping Automated Endothelial Keratoplasty (DSAEK), lamellar keratoplasty)
  * Previous anterior or posterior chamber surgery (e.g., vitrectomy, laser iridotomy)
  * Moderate-to-advanced glaucoma
  * Strabismus
  * Use of arcuate incisions for astigmatism management at the time of surgery
  * Diabetic retinopathy
  * Macular pathology (e.g. age-related macular degeneration, epiretinal membrane, etc.)
  * History of retinal detachment
  * Subjects who have an acute or chronic disease or illness that would confound the results of this investigation (e.g., immunocompromised, connective tissue disease, clinically significant atopic disease, diabetes, and any other such disease or illness), that are known to affect postoperative visual acuity.
  * Participation in (or current participation) any investigational drug or device trial within the previous 30 days prior to the start date of this trial.

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2018-10-05 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clayton G Blehm, MD, Principal Investigator — Gainesville Eye Associates
Locations (1):
- Gainesville Eye Associates, Gainesville, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ReSTOR Toric
Started | 29
Completed | 29
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | ReSTOR Toric
Number analyzed (Participants) | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Residual Refractive Cylinder
Description: Manifest postoperative refractive cylinder (measured in diopters, with a phoropter or trial lens set) after cataract surgery and IOL implantation
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: diopters
Arm/Group | ReSTOR Toric
Number analyzed (Participants) | 29
diopters | 0.02 (0.08)

2. Secondary Outcome: Monocular Uncorrected Near Visual Acuity
Description: Monocular uncorrected near visual acuity measuring in logMAR
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Toric
Number analyzed (Participants) | 29
logMAR | 0.12 (0.11)

3. Secondary Outcome: Monocular Uncorrected Distance Visual Acuity
Description: Monocular uncorrected distance visual acuity measured in logMAR notation
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Toric
Number analyzed (Participants) | 29
logMAR | 0.04 (0.09)

4. Secondary Outcome: Monocular Uncorrected Intermediate Visual Acuity
Description: Monocular Uncorrected intermediate visual acuity measured in logMAR notation (log of the minimum angle of resolution)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Toric
Number analyzed (Participants) | 29
logMAR | 0.06 (0.11)

5. Secondary Outcome: Monocular Best Corrected Distance Visual Acuity
Description: Monocular best corrected distance visual acuity measured in logMAR notation
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Toric
Number analyzed (Participants) | 29
logMAR | .04 (.09)

6. Secondary Outcome: Monocular Best Distance-corrected Intermediate Visual Acuity
Description: Monocular best distance-corrected intermediate visual acuity in logMAR notation
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Toric
Number analyzed (Participants) | 29
logMAR | .06 (.11)

7. Secondary Outcome: Monocular Best Distance-corrected Near Visual Acuity
Description: Monocular best distance-corrected near visual acuity measured in logMAR notation
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Toric
Number analyzed (Participants) | 29
logMAR | .11 (0.12)

8. Secondary Outcome: Binocular Uncorrected Near Visual Acuity
Description: Binocular uncorrected near (40cm) visual acuity measured in logMAR notation
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Toric
Number analyzed (Participants) | 29
logMAR | 0.01 (0.08)

9. Secondary Outcome: Binocular Uncorrected Distance Visual Acuity
Description: Binocular uncorrected distance visual acuity measured in logMAR notation
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Toric
Number analyzed (Participants) | 29
logMAR | -0.01 (0.07)

10. Secondary Outcome: Binocular Uncorrected Intermediate Visual Acuity
Description: Binocular uncorrected intermediate (60cm) visual acuity
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Toric
Number analyzed (Participants) | 29
logMAR | -0.02 (0.07)

11. Secondary Outcome: Binocular Best-corrected Distance Visual Acuity
Description: Binocular best-corrected distance visual acuity measured in logMAR notation
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Toric
Number analyzed (Participants) | 29
logMAR | -0.03 (0.05)

12. Secondary Outcome: Binocular Best Distance-corrected Intermediate Visual Acuity
Description: Binocular best distance-corrected intermediate (60cm) visual acuity
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Toric
Number analyzed (Participants) | 29
logMAR | -0.06 (0.03)

13. Secondary Outcome: Binocular Best Distance-corrected Near Visual Acuity
Description: Binocular best distance-corrected near (40cm) visual acuity
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Toric
Number analyzed (Participants) | 29
logMAR | 0.01 (0.01)

14. Secondary Outcome: IOL Orientation
Description: Postoperative orientation changes with the Toric ReSTOR IOL up to 3 months after surgery will be measured by determining the angle of orientation of the IOL in degrees (0-180) using a slit lamp.
Time Frame: 3 months
Population: Subjects are enrolled, eyes (2x subjects) were evaluated for some tests.
Measure: Number; unit: Eyes with < 5 degrees rot'n from 1-3 mos
Units Other Than Participants: Eyes
Arm/Group | ReSTOR Toric
Number analyzed (Participants) | 29
Number analyzed (Eyes) | 58
Eyes with < 5 degrees rot'n from 1-3 mos | 56

15. Secondary Outcome: Binocular Best Distance-corrected Defocus Curve
Description: Binocular best distance-corrected defocus curve.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR Acuity
Arm/Group | ReSTOR Toric
Number analyzed (Participants) | 29
logMAR Acuity
  Defocus +1.00 | .24 (.20)
  Defocus +0.50 | .07 (.11)
  Defocus 0.00 | -.01 (0.07)
  Defocus -4.00 | .55 (.19)
  Defocus -3.50 | .40 (.15)
  Defocus -3.00 | .28 (.12)
  Defocus -2.50 | .19 (.11)
  Defocus -2.00 | .16 (.11)
  Defocus -1.50 | .21 (.11)
  Defocus -1.00 | .19 (.08)
  Defocus -0.50 | 0.08 (0.10)

16. Secondary Outcome: Binocular Uncorrected Defocus Curve.
Description: Binocular uncorrected defocus curve, from +1.0D to -4.00D in 0.50D increments
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: logMAR Acuity
Arm/Group | ReSTOR Toric
Number analyzed (Participants) | 27
logMAR Acuity
  Defocus 1.00 | .22 (.20)
  Defocus 0.50 | .07 (.11)
  Defocus 0.00 | -.01 (.08)
  Defocus -4.00 | .55 (.19)
  Defocus -3.50 | .41 (.16)
  Defocus -3.00 | .29 (0.13)
  Defocus -2.50 | .18 (.11)
  Defocus -2.00 | .16 (.11)
  Defocus -1.50 | .20 (.11)
  Defocus -1.00 | .19 (.08)
  Defocus -0.50 | 0.09 (.10)

17. Secondary Outcome: Subjective Visual Quality
Description: Quality of vision, measured with a subjective questionnaire (Q of V). Frequency, Severity and "Degree of Bother" aggregate statistics. Scored on a Rasch scale (0-100) where lower is better.
Time Frame: 3 months
Measure: Median (Full Range); unit: score on a Rasch scale (0-100)
Arm/Group | ReSTOR Toric
Number analyzed (Participants) | 29
score on a Rasch scale (0-100)
  Frequency | 32 [0 to 72]
  Severity | 22 [0 to 54]
  Degree of Bother | 0 [0 to 60]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | ReSTOR Toric
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT03856944/Prot_SAP_001.pdf